CLINICAL TRIAL: NCT04123015
Title: Clinical Activity During Night-shift: an Ecological Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pauline Darbellay Farhoumand, Principal Investigator, University Hospital, Geneva
Other Study IDs: SMIG_001
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Nightshift Work; Handoff Sessions; Stress, Psychological; Regret; Sleep
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A convenient sample of internal medicine residents will be observed during their nightshift work in the wards of the department of internal medicine of a university hospital. The epidemiology of night calls and emergencies, including incidence, causes, management, and prognosis, will be assessed prospectively. The impact of nightshift work on sleep, stress, quality of life, regrets, and general well being of the residents observed will be measured through completion of validated questionnaires. Quality of handoff sessions will also be assessed.

DETAILED DESCRIPTION:
Various medical problems of patients admitted to an internal medicine ward can worsen during the stay. Furthermore, new, unidentified problems can develop (complications, medication errors, delirium, acute anxiety or pain, etc). During evenings, nights and week-ends, emergent needs of hospitalized patients are usually cared for by physicians in-training, who are in charge of a large number of patients. Hence, physicians should have a wide range of medical knowledge and procedural skills and know how acute problems are dealt with in the unique environment of the healthcare institution. Training physicians should also be able to obtain information and counseling efficiently, either from clinical guidelines, senior supervisors, or specialists.

These requirements may represent a significant stress for training physicians and may have a major impact on their health, quality of life, and finally on the quality of inpatient care. Nightshift work may lead later to a high burden of regrets among caregivers.

Better knowledge of training needs, organization features, coping strategies, and regrets associated with nightshift duty are important to prepare training physicians to that demanding and necessary task. Understanding of the epidemiology of night-shift ward emergencies could provide guidance concerning the required level of staffing and training of the responding medical team.

Furthermore, efficient transmission of information between day and night staff (so-called handoffs) is a difficult yet important part of care. Systematic observation of handoff sessions between physicians before and after nightshifts may enhance previous knowledge on key components of these topics.

The investigators will evaluate the incidence causes, and prognosis of night-shift emergencies in internal medicine wards by direct observation of the nightshift work of a convenient sample of internal medicine residents. By the means of before-and-after shift completion of various validated questionnaires, the investigators will explore quantitatively and qualitatively the physiological and psychological impact on nightshift work for physicians in training.

The planned study will also provide qualitative and quantitative data concerning handoffs session, and the repercussions on night shift emergencies management.

ELIGIBILITY:
Inclusion Criteria:

* resident in training in the internal medicine department, involved in one or more nightshift during the study

Exclusion Criteria:

* unwilling to participate

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: see above
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Incidence of nightshift interventions | 12 hours
% of patients with nightshift interventions of different intensity | 12 hours
  Rated on an ad-hoc scale (from "phone intervention only" to "active resuscitation")
% of patients with different causes of nightshift interventions | 12 hours
  Rated on an ad-hoc scale listing the different causes (e.g. acute confusion; chest pain, etc)
Incidence of selected outcomes of nightshift intervention | 24 hours
  Rated on an ad-hoc scale (from "death" to "problem resolves without further intervention"
Incidence of specific interventions during nightshift | 12 hours
  Rated on an ad-hoc list, from "Provision of CPR or intubation" to "Prescription of any new drug"
Incidence of predictable nightshift emergencies | 12 hours
  Rated on an ad-hoc scale, from "Unexpected" to "Expected"
Incidence of preventable nightshift emergencies | 12 hours
  Rated on an ad-hoc scale, from "Unpreventable" to "Very likely preventable"

SECONDARY OUTCOMES:
incidence of sleep problems in nightshift residents | 30 days
severity of sleep problems in nightshift residents | 30 days
  measured with the insomnia severity index questionnaire, ISI
incidence of stress symptoms in nightshift residents | 30 days
severity of stress symptoms in nightshift residents | 30 days
  Measured with an ad hoc scale (From "no stress at all" to "intense stress most of the time")
incidence of regrets in nightshift residents | 30 days
severity of regrets in nightshift residents | 30 days
  Measured with the regret intensity questionnaire(RIS-10)
incidence of burnout symptoms in nightshift residents | 30 days
severity of burnout symptoms in nightshift residents | 30 days
  Measured with the Copenhagen Burnout Inventory, CBI

CONTACTS AND LOCATIONS:
Overall Officials: Pauline DARBELLAY FARHOUMAND, MD, Principal Investigator — Geneva University Hospitals, General Internal Medicine Department
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland